CLINICAL TRIAL: NCT04106024
Title: Efficacy and Safety of Anlotinib in Patients With Advanced Gastrointestinal Stromal Tumor After Failure of Imatinib: a Prospective, Single Arm and Multicenter Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cttq (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018YJZ42
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 12mg.qd ,taken for 2 weeks and discontinued for 1 week, namely 3 weeks (21 days).

SUMMARY:
Gastrointestinal stromal tumors (GIST) compose approximately 20% of soft tissue sarcomas with an annual incidence of approximately 7 per million population. GISTs occur throughout the GI tract, most commonly in the stomach or small intestine. The main treatment for localised GIST is surgical resection. At least 40% of these patients will develop recurrence or metastasis following complete resection. Local recurrence, liver metastases and/or dissemination within the abdominal cavity are the most common clinical manifestations. Although imatinib and sunitinib has greatly improved the quality of life and survival of patients with advanced GIST. Analysis of clinical trials revealed that patients with tumours with KIT exon 17 or 18 mutations, with a second mutation in KIT exon 17 or 18, had worse responses to imatinib and sunitinib. Some patients with PDGFRA D842V mutation do not respond to the present standard therapies.

Anlotinib (1-[[[4-(4-fluoro-2-methyl-1H-indol-5-yloxy)-6-methoxyquinolin-7-Yl] oxy] methyl]cyclopropanamine dihydrochloride) , a multi-targeted tyrosine kinase inhibitor (TKI), characterized as a highly selective and potent c-KIT, VEGFR, PDGFR, FGFR inhibitor. In vitro and in vivo, Anlotinib has a broad spectrum of inhibitory action on tumor angiogenesis and growth, which showed broad activity against soft tissue sarcoma and GIST with D842V, D816H, V560G and V654A mutations. In 2015, the US FDA granted orphan drug treatment for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

- 1. Male or female, 18 years of age or older. 2. Histologically-proven diagnosis of recurrent or metastatic GIST (Gastrointestinal Stromal Tumors).

3. Patients must have measurable disease meeting the requirement of RECIST 1.1. 4. Failure of prior treatment with imatinib or intolerant to imatinib. 5. No condition for receiving sunitinib and regorafenib. 6. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1. Resolution of all acute toxic effects Adequate organ function. 7. The estimated survival period is more than 3 months. 8. Ability to understand and the willingness to sign a written informed consent document 9. Subject will comply with the study procedures and therapy

Exclusion Criteria:

* 1. Local or metastatic GIST is resectable. 2. Be treated with sunitinib or regorafenib. 3. AST and/or ALT > 2.5 times ULN, or Bilirubin >1.5 times upper limit of normal (ULN) 4. Neutrophil count < 1.5 x 10^9/L, or Platelet count <75 x 10^9/L, or Hemoglobin<90g/L 5. Cr >1.5×ULN 6. Other malignancy within the past 5 years except for adequately treated carcinoma in situ of the cervix or cutaneous basal cell carcinoma.

  7. Known brain metastasis, spinal cord compression, carcinomatous meningitis, or cerebral or soft meningeal disease through CT or MRI during screening stage.

  8. Within the past 1 years, subjects have one of the following disease: myocardial infarction, serious/instable angina pectoris, symptomatic congestive heart failure or cerebrovascular accident from coronary/peripheral artery bypass grafting.

  9. Known human immunodeficiency virus positivity. 10. Joining in other trail. 11. Women who are pregnant or lactating; No contraception for subject during childbearing period.

  12. Subject with other serious acute and chronic physical or mental problems, or laboratory abnormality, will increase the risks associated with trail or drug. It will also interference the judgment of the results. In the judgment of the investigator, subject is inadequate to participant the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 18 month
  Progress Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wu, Principal Investigator — Chinese PLA General Hospital; Xinhua Zhang, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Ye Zhou, Principal Investigator — Fudan University; Bo Zhang, Principal Investigator — West China Hospital; XiaoFeng Sun, Principal Investigator — Jiangsu Cancer Institute & Hospital; HongYan Qu, Principal Investigator — Harbin Medical University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China